CLINICAL TRIAL: NCT04817488
Title: Live Stream of Prehospital Emergency Ultrasound in Patients With Acute Dyspnoea
Status: Active, not recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christina Hafner, Clinical Investigator, Medical University of Vienna
Other Study IDs: 2411/2020
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Echocardiography; Acute Dyspnea
Keywords: Ultrasound diagnostics; Prehospital emergency medicine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prehospital emergency ultrasound with tele-supervision: Prehospital emergency ultrasound of patients with acute dyspnea will be performed with tele-supervision.
  Interventions: Other: Prehospital emergency ultrasound with tele-supervision
- Prehospital emergency ultrasound without tele-supervision: Prehospital emergency ultrasound of patients with acute dyspnea will be performed without tele-supervision.
  Interventions: Other: Prehospital emergency ultrasound without tele-supervision

INTERVENTIONS:
Other: Prehospital emergency ultrasound with tele-supervision — Prehospital emergency ultrasound with tele-supervision in patients with acute dyspnoea
  Groups: Prehospital emergency ultrasound with tele-supervision
Other: Prehospital emergency ultrasound without tele-supervision — Prehospital emergency ultrasound without tele-supervision in patients with acute dyspnoea
  Groups: Prehospital emergency ultrasound without tele-supervision

SUMMARY:
Background: Acute dyspnoea is a common symptom in prehospital emergency medicine. As ultrasound gained in importance for diagnosis in patients with acute respiratory distress, it plays even a role in the prehospital setting. However, prehospital emergency ultrasound (PEU) remains challenging and requires knowledge and skills. New prehospital ultrasound devices offer the possibility for tele-supervision. The impact of tele-supervision of PEU in patients with acute dyspnoea is unclear.

Objective: This prospective observational study aims to evaluate the effect of PEU with tele-supervision on diagnosis, treatment strategies and cognitive load in comparison to PEU without tele-supervision in patients with acute dyspnoea.

Methods: In total 350 prehospital emergency patients with acute dyspnoea will be included in this study. Patients will be observed in two groups. In group 1 PEU will be performed with tele-supervision, whereas in group 2 PEU will be performed without tele-supervision (tele-supervision not available).

ELIGIBILITY:
Inclusion Criteria:

Patients will be included, if they suffer from acute dyspnoea and at least one of the two following signs of respiratory failure:

* Respiratory rate >20 breaths per minute
* Peripheral oxygen saturation without oxygen supplementation <90%

Exclusion Criteria:

* under the age of 18
* if PEU will lead to a delay of live-saving treatment or transportation
* if patient rejects the PEU, the patient will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 350 critically ill patients with acute dyspnoea will be included in this study. In 175 patients ultrasound with tele-supervision and in 175 patients ultrasound without tele-supervision will be performed. Allocation to one of the two groups depends on the availability of tele-supervision. Tele-supervision is available in 50% of the time.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of prehospital diagnosis after PEU in relation to the (correct) in-hospital diagnosis | through study completion, an average of 1 year
  The aim of this study is to compare the accuracy of a prehospital emergency ultrasound (PEU) done with or without tele-supervison in patients suffering from acute dyspnoea and evaluate the accuracy of the diagnosis in relation to the (correct) in-hospital diagnosis.

SECONDARY OUTCOMES:
Agreement of diagnosis before PEU and after PEU | through study completion, an average of 1 year
  Is there an agreement between the diagnosis before performing the prehospital emergency ultrasound (PEU) and after performing it.
Duration of prehospital emergency ultrasound (PEU) | through study completion, an average of 1 year
  Duration of prehospital emergency ultrasound (PEU)

CONTACTS AND LOCATIONS:
Overall Officials: Department of Anaesthesia & General Intensive Care, Study Chair — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Department of Anaesthesia & General Intensive Care, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided